CLINICAL TRIAL: NCT06747780
Title: Text Messaging Intervention on Happy Family Meal for Improving Family Communication and Well-being in Hong Kong Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Wang Man-Ping (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Sponsor-Investigator, Dr. Wang Man-Ping, Prof, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: JCSFLP2-TMI
Record Dates: First submitted 2024-12-12; First posted 2024-12-24 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: N/A - Healthy Subjects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Participants and their eligible family members in the intervention group will receive a digital booklet via MMS and daily text messages related to happy family meals via SMS for two weeks. The content of these messages will be based on five positive psychology themes: joy, gratitude, flow, savoring, and listening, adapted from the Happy Family Kitchen II project. Participants in the intervention group will receive notifications prompting them to join two family-based activities, adapted from the Happy Family Kitchen II project, as boosters at one-month and three-month after they receive the daily SMS, respectively.
  Interventions: Behavioral: Text messaging
- Waitlist control group (Other): Participants in the waitlist control group will not receive the intervention immediately but will be offered the same 14-day SMS intervention and two family-based activities three months post-intervention.
  Interventions: Behavioral: Control (Usual care)

INTERVENTIONS:
Behavioral: Text messaging — A digital booklet, text messages for two weeks, and two family-based activity boosters
  Arms: Intervention group
Behavioral: Control (Usual care) — Control only
  Arms: Waitlist control group

SUMMARY:
Family meals are crucial for family communication and well-being. This text messaging intervention digitalizes Happy Family Kitchen II, a face-to-face community-based intervention previously shown to be effective.

This is a two-arm, parallel-group, randomized controlled trial (RCT) designed to evaluate the effectiveness of a text messaging intervention aimed at promoting happy family meals among Hong Kong adults. Eligible participants are Hong Kong residents aged 18 or older, with at least one parent or child also aged 18 or older, who can read Chinese and have access to Short Message Service (SMS) and Multimedia Messaging Service (MMS) platforms. A target of approximately 1,050 participants will be stratified by four types of family roles and negative emotional eating status and randomized to either the intervention group, receiving a digital booklet, text messages for two weeks, and two family-based activity boosters, or the waitlist control group. The content is based on five positive psychology themes: joy, gratitude, flow, savoring, and listening. Primary outcomes include improvement in family communication and well-being at three months post-intervention.

This study aims to assess the effectiveness of a digital intervention on family communication and well-being through the promotion of happy family meals. By leveraging information communication technologies (ICTs), this intervention offers a scalable and cost-effective approach, providing insights into the feasibility and effectiveness of digitizing community-based interventions.

DETAILED DESCRIPTION:
Background:

Family meals are a cornerstone of family communication and well-being. Studies have shown that the benefits of quality family meals include not only nutritional intake but also improved family well-being (family health, happiness, harmony, i.e., the family 3Hs), with family communication quality playing a pivotal role. Urban lifestyles limit opportunities for family communication and gatherings, which are crucial to family bonding. Surveys have shown that Chinese individuals rarely heed their parents' advice on important matters and lack knowledge on positive family communication.

Information communication technologies (ICTs) diversify modes of family communication and offer intriguing opportunities to promote family communication and well-being. Leveraging ICTs in brief behavioral interventions can be impactful in influencing decision-making. Text messaging interventions have shown promise in smoking cessation, weight management, and medication adherence. Text messaging via SMS can provide practical suggestions for positive family communication and encourage participation in family meals with tailored messages specific to challenges faced by Hong Kong families, such as time constraints and conflicting schedules. Evidence from similar ICT-based interventions supports the potential effectiveness of text messaging in promoting family meals as a ubiquitous and easy-to-use medium. A randomized controlled trial (RCT) by Patrick et al. showed that text message reminders significantly improved dietary habits and meal planning among participants. A study by Fulkerson et al. showed that a web-based intervention for family meals led to increased family meal frequency and improved dietary outcomes.

Happy Family Kitchen (HFK I), Happy Family Kitchen II (HFK II), and Happy Family Kitchen Movement (HFKM) were community-based interventions under The FAMILY Project, which highlighted the effectiveness of face-to-face cooking and dining activities in improving family communication and well-being. As part of The Jockey Club SMART Family-Link Project, the investigators aim to digitalize the Happy Family Kitchen initiative with the framework of five positive psychology themes: joy, gratitude, flow, savoring, and listening, providing a cost-effective and scalable approach. This trial aims to evaluate the effectiveness of a text messaging intervention on happy family meals for improving family communication and well-being in Hong Kong adults.

Hypothesis:

Higher scores in the family communication scale and family well-being for participants in the intervention group than the waitlist control group at three-month post-intervention.

Study Design:

This study is a two-arm, parallel-group, randomized controlled trial (RCT) aimed at evaluating the effectiveness of a text messaging intervention on promoting happy family meals to improve family communication and well-being among Hong Kong adults.

Randomization and Blinding:

Participants who meet the inclusion criteria will be randomly assigned to either the intervention group or the waitlist control group in a 1:1 ratio using computer-generated random numbers. The randomization will be stratified based on the Chinese Version of the Weight-Related Eating Questionnaire - Emotional Eating subscale (WREQ-EE) and four types of family roles:

1. Children of the family aged 18 or above (whether living with parents or not, no children).
2. Parents with children of the family under 18 years old.
3. Parents with children of the family aged 18 or above (unmarried or living with parents).
4. Parents with children of the family aged 18 or above (married or living independently).

The allocation concealment will be maintained by the researchers involved in recruitment and implementation, who will generate the list of participants completing the baseline questionnaire for randomization. Blinding will be applied to the data analysts and the participants.

Intervention Group:

Participants and their eligible family members in the intervention group will receive a digital booklet via MMS and daily text messages related to happy family meals via SMS for two weeks. The content of these messages will be based on five positive psychology themes: joy, gratitude, flow, savoring, and listening, adapted from the Happy Family Kitchen II project. Participants in the intervention group will receive notifications prompting them to join two family-based activities, adapted from the Happy Family Kitchen II project, as boosters at one-month and three-month after they receive the daily SMS, respectively.

Control Group:

Participants in the waitlist control group will not receive the intervention immediately but will be offered the same digital booklet, 14-day SMS intervention and two family-based activities boosters at three months post-intervention.

ELIGIBILITY:
Inclusion criteria:

1. are Hong Kong adults aged 18+ years who have at least one parent or children (aged 18+ years) other than their spouse in the family,
2. can read Chinese,
3. have access to SMS/MMS platform, and
4. give informed consent (team leaders only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in family communication | Baseline, 3-month post-intervention
  Family communication will be assessed using the 10-item Family Communication Scale, which measures satisfaction with family communication, listening skills, expression of affection, and problem-solving abilities. Responses are scored on a five-point scale from 1 to 5, with total score ranging from 10 to 50 and higher scores indicating better communication.
Changes in family well-being | Baseline, 3-month post-intervention
  Family well-being will be measured using three separate questions: "Do you think your family is harmonious/happy/healthy?", each asking respondents to rate their family health, happiness, or harmony on a scale from 0 to 10, with higher scores indicating better outcomes.

SECONDARY OUTCOMES:
Changes in family communication | Baseline, 1-month post-intervention
  Family communication will be assessed using the 10-item Family Communication Scale, which measures satisfaction with family communication, listening skills, expression of affection, and problem-solving abilities. Responses are scored on a five-point scale from 1 to 5, with higher scores indicating better communication, with total score ranging from 10 to 50 and higher scores indicating better communication.
Changes in family well-being | Baseline, 1-month post-intervention
  Family well-being will be measured using three separate questions: "Do you think your family is harmonious/happy/healthy?", each asking respondents to rate their family health, happiness, or harmony on a scale from 0 to 10, with higher scores indicating better outcomes.
Changes in family meal behavioral outcomes | Baseline, 1-month post-intervention and 3-month post-intervention
  Family meal behavioral outcomes will be measured using the duration of meals (minutes per meal) and the frequency of five positive psychology experiences (times per week) in the past 7 days.
Changes in symptoms of anxiety and depression | Baseline, 1-month post-intervention and 3-month post-intervention
  Symptoms of anxiety and depression will be assessed using the Patient Health Questionnaire-4 (PHQ-4). Respondents will indicate the frequency of the described symptoms over the previous two weeks using a 4-point Likert scale from 0 (not at all) to 3 (nearly every day). The total score of each subscale ranges from 0 to 6, with higher scores indicating worse outcomes.
Changes in personal happiness | Baseline, 1-month post-intervention and 3-month post-intervention
  Personal happiness will be measured by asking, "How happy do you think you are?" with responses from 0 (very unhappy) to 10 (very happy).
Changes in personal xingfu | Baseline, 1-month post-intervention and 3-month post-intervention
  Personal xingfu will be measured by asking, 'How xingfu do you think you are?' with responses from 0 to 10 and higher score indicating better personal xingfu.
Changes in family xingfu | Baseline, 1-month post-intervention and 3-month post-intervention
  Family xingfu will be measured by asking, 'How xingfu do you think your family xingfu is?' with responses from 0 to 10 and higher score indicating better family xingfu.
Changes in family communication quality | Baseline, 1-month post-intervention and 3-month post-intervention
  Family communication quality will be measured by having respondents rate the quality of communication between themselves and their family members on an 11-point scale (0-10), with higher scores indicating better family communication quality.
Changes in healthiness of diet | Baseline, 1-month post-intervention and 3-month post-intervention
  The healthiness of the diet will be measured by respondents rating their diet healthiness on an 11-point scale (0-10), with higher scores indicating healthier diet.
Changes in physical activity | Baseline, 1-month post-intervention and 3-month post-intervention
  Physical activity will be measured by having respondents rate their physical activity on an 11-point scale (0-10), with higher scores indicating more sufficient physical activity.
Changes in Weight-Related Eating Questionnaire - Emotional Eating subscale | Baseline, 1-month post-intervention and 3-month post-intervention
  The Weight-Related Eating Questionnaire Emotional Eating subscale (WREQ-EE) will be used to assess emotional eating on a scale of 1 to 5, with total scores ranging from 4 to 20 and higher scores indicating worse emotional eating.
Process evaluation | 1-month post-intervention and 3-month post-intervention
  Process evaluation will be measured using a perceived benefits question, an assessment of whether the messages were read, and by asking respondents to rate the importance, confidence, and difficulty of happy family meal on 11-point scales (0-10), with higher score indicating better outcomes.

IPD SHARING:
Plan to Share IPD: No